CLINICAL TRIAL: NCT06392620
Title: Effects of Telerehabilitation in Patients With Ankylosing Spondylitis
Brief Title: Telerehabilitation in Ankylosing Spondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/03-08
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondilitis,; Exercise; YouTube
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): An individually planned exercise program including stretching, strengthening, respiratory, aerobic and posture exercises will be applied via video conference method.
  Interventions: Other: Study Group
- Control group (Experimental): It will be recommended a video on YouTube platform and will be asked to do the exercises by following the content of these videos
  Interventions: Other: Study Group

INTERVENTIONS:
Other: Study Group — n individually planned exercise program including stretching, strengthening, respiratory, aerobic and posture exercises will be applied via video conference method

SUMMARY:
Ankylosing Spondylitis (AS) is an inflammatory rheumatic disease primarily affecting the spine and sacroiliac joint. xercise is one of the most important nonpharmacologic treatment modalities in AS. Stretching, strengthening, aerobic, posture, balance and moltimodal exercise methods are the most commonly used treatment methods. The study will include 44 patients diagnosed with AS aged 18-65 years. Patients will be divided into two randomized controlled groups with 22 patients in each group. Group 1 will receive a personalized exercise program including stretching, strengthening, respiratory, aerobic and posture exercises via video conferencing. Group 2 will be recommended a video on the YouTube platform and will be asked to perform the exercises by following the content of these videos. Spinal mobility will be assessed with Bath Ankylosing Spondylitis Metrology Index, disease activity with Bath Ankylosing Spondylitis Disease Activity Index, function with Bath Ankylosing Spondylitis Function Index, quality of life with Ankylosing Spondylitis Quality of Life Scale and posture with PostureScreeen mobile application.

DETAILED DESCRIPTION:
Ankylosing Spondylitis (AS) is an inflammatory rheumatic disease primarily affecting the spine and sacroiliac joint. It usually begins in the second decade of life and is more common in men than women. The benefits of exercise and physical activity in health and disease are well recognized. Exercise is one of the most important nonpharmacologic treatment modalities in AS. Stretching, strengthening, aerobic, posture, balance and moltimodal exercise methods are the most commonly used treatment modalities. However, the application of these exercise methods to patients with AS in the form of a home exercise program is advantageous due to its low cost and the ease with which patients can start exercising. The study will include 44 patients diagnosed with AS aged 18-65 years. Patients will be divided into two randomized controlled groups with 22 patients in each group. Group 1 will receive a personalized exercise program including stretching, strengthening, respiratory, aerobic and posture exercises via video conferencing. Group 2 will be recommended a video on the YouTube platform and will be asked to perform the exercises by following the content of these videos. Patients in Group 2 will be followed up by regular communication with the patients and by asking the patient to create an attendance chart. Patients in both groups will receive the treatment 3 days a week for 8 weeks. Evaluation methods will be applied at the beginning and at the end of the treatment. Spinal mobility will be assessed with Bath Ankylosing Spondylitis Metrology Index, disease activity with Bath Ankylosing Spondylitis Disease Activity Index, function with Bath Ankylosing Spondylitis Function Index, quality of life with Ankylosing Spondylitis Quality of Life Scale and posture with PostureScreeen mobile application.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Patients whose medical treatment has not changed in the last three months
* Patients with a diagnosis of AS will be included.

Exclusion Criteria:

* Patients who are pregnant
* Patients with a diagnosis of malignancy
* Patients with other concomitant systemic inflammatory rheumatic diseases
* Patients with neurological, orthopedic or congenital problems that prevent physical activity
* Patients with regular exercise habits will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Spinal mobility | 10 minutes
  Spinal mobility will be assessed and scored with BASMI. According to the index, there are five measurements: lateral lumbar flexion, tragus-wall distance, lumbar flexion (Modified Schober), maximal intermalleolar distance and cervical rotation.

SECONDARY OUTCOMES:
Disease activity | 1 minute
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) consisting of 6 questions will be used to assess disease activity.
Function | 2 minutes
  BASFI will be used to assess function. The index includes 10 questions about activities of daily living. A 10 cm VAS will be used for each question

CONTACTS AND LOCATIONS:
Overall Officials: Songul Baglan Yentur, Principal Investigator — Firat University
Locations (1):
- Songul Baglan Yentur, Elâzığ, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yentur SB, Boyrazli IS, Elbasti MS, Koca SS. Effects of telerehabilitation and YouTube platform-based exercise videos in patients with axial spondyloarthritis: a randomized controlled study. Clin Rheumatol. 2025 Sep;44(9):3561-3571. doi: 10.1007/s10067-025-07591-w. Epub 2025 Jul 25. PMID 40715923